CLINICAL TRIAL: NCT02506127
Title: A Sham-controlled Study of Prefrontal Intermittent Theta Burst Stimulation in Major Depressive Disorder
Brief Title: Intermittent Theta Burst Stimulation for MDD
Acronym: iTBS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol discontinued for futility
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-000701
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: TBS, MDD, Sham-controlled, neuromodulation, TMS
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open-label (Experimental): Theta burst stimulation (TBS) is a form of repetitive transcranial magnetic stimulation (TMS). Standard TBS parameters consisting of 3-pulse, 50Hz bursts every 200 ms (5 Hz) at an intensity of 80% motor threshold (MT) will be utilized. Intermittent TBS will be delivered in 2-second trains of bursts repeated every 10 seconds for a total of 570 seconds (1800 pulses) in each session.
  Each treatment session thus involves < 10 minutes of stimulation. The subject and researchers know what treatment is being administered.
  Interventions: Device: Neuronetics XPLOR system
- Blinded Active (Active Comparator): Standard TBS parameters consisting of 3-pulse, 50Hz bursts every 200 ms (5 Hz) at an intensity of 80% motor threshold (MT) will be utilized. Intermittent TBS will be delivered in 2-second trains of bursts repeated every 10 seconds for a total of 570 seconds (1800 pulses) in each session.
  Each treatment session thus involves < 10 minutes of stimulation. The subject and researcher will not know what type of treatment will be administered.
  Interventions: Device: Neuronetics XPLOR system
- Blinded Sham (Sham Comparator): This is a sham treatment which will mimic the open-label and blinded active to enable the effects of the supposedly "active" treatment to be assessed objectively. The subject and researcher will not know what type of treatment will be administered.
  Each treatment session will be < 10 minutes in duration.
  Interventions: Device: Neuronetics XPLOR system

INTERVENTIONS:
Device: Neuronetics XPLOR system — Transcranial magnetic stimulation system

SUMMARY:
This study will evaluate the effectiveness of intermittent Theta Burst Stimulation for patients with Major Depressive Disorder.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate the effectiveness and efficacy of intermittent Theta Burst Stimulation (iTBS) for treatment of Major Depressive Disorder (MDD). Subjects will be randomly assigned to two weeks (10 sessions) of treatment with open-label iTBS, blinded iTBS or blinded sham. 'Open-label' means that you (the subject) and the study staff will know that you are receiving active iTBS treatment. 'Blinded' or 'sham-controlled' means that you, the subject, will not know whether the treatment you receive is the active treatment or the non-active treatment. In the 'sham' condition, the stimulator will turn on but will not actually be stimulating your brain. Subjects who do not show remission of symptoms after the first 2 weeks of treatment will receive 10 additional treatment sessions with open-label active iTBS. Subjects will be evaluated at Week 12 to assess the durability of symptoms changes.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with non-psychotic, unipolar Major Depressive Disorder (MDD) assessed via the MINI structured interview
2. Must have been on a stable dose of antidepressant medication (excluding tricyclic antidepressants) for at least 1 month prior to randomization, and with significant residual MDD symptoms as evidenced by a HamD17 score > 17;
3. If receiving medication other than for depression (e.g., anxiety, sleep, mood stabilization), must have been on stable dose for at least 1 month prior to randomization
4. A history of treatment failure with at least one adequate trial of an antidepressant medication in the current episode, assessed by the Antidepressant Treatment and History Form
5. Age range: 22-65.

Exclusion Criteria:

1. Patient is mentally or legally incapacitated, unable to give informed consent.
2. Patients with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime)); bipolar disorder (lifetime); dementia (lifetime); current Mini Mental State Examination ≤ 24; delirium or substance abuse within the past 6 months; eating disorder within the past year; obsessive-compulsive disorder (lifetime); post-traumatic stress disorder within the past year; acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
3. Patients with a HamD suicidality item score of '3' or '4,' corresponding to "suicidal ideas or gestures" or "attempts at suicide," will be excluded.
4. Patients with exposure to Electroconvulsive Therapy within the past 6 months, previous TMS treatment for any condition, or Vagus Nerve Stimulation treatment (lifetime).
5. Patients who have met diagnostic criteria for any current substance abuse disorder at any time in the 6 months prior to enrollment.
6. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, Cerebral Vascular Accident, or Transient Ischemic Attacks; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
7. Any history of intracranial implant including cochlear implant, implanted electrodes/stimulators, aneursym clips or coils, stents, bullet fragments; implanted cardiac pacemaker, defibrillator, vagus nerve stimulator, deep brain stimulator; or other implanted devices or objects contraindicated by product labeling.
8. Neurological conditions including epilepsy, cerebrovascular disease, dementia, increased intracranial pressure, history of repetitive or severe head trauma, or with primary or secondary tumors in the Central Nervous System.
9. current pregnancy, breast feeding, or not using a medically accepted means of contraception.
10. Infection or loss of integrity of skin over the forehead, where the device will be positioned.
11. Increased risk of seizure as indicated by: a) history (or family history) of seizure or epilepsy; b) history of stroke, head injury, or unexplained seizures; c) concurrent medication use such as tricyclic antidepressants, neuroleptic medications, or other drugs that are known to lower the seizure threshold; d) secondary conditions that may significantly alter electrolyte balance or lower seizure threshold; e) no quantifiable motor threshold such that TMS dosage cannot be accurately determined.
12. Other medical contraindications to any of the study procedures.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-09 (Actual); Primary Completion 2027-12-08 (Estimated); Study Completion 2027-12-08 (Estimated)

PRIMARY OUTCOMES:
Percent change in Hamilton Depression Scale (HamD17) | two week

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA TMS Clinic and Research Service, Los Angeles, California, United States